CLINICAL TRIAL: NCT03494608
Title: Evaluation of Postoperative Cognitive Function, Anxiety, Depression and Quality of Life in Patients With Unruptured Intracranial Aneurysms: a Multi-center Prospective Cohort Study
Brief Title: Evaluation of Postoperative Cognitive Function, Anxiety, Depression and Quality of Life in Patients With Unruptured Intracranial Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: West China Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief nurse of Neurosurgery Department, professor, Xuanwu Hospital, Beijing
Other Study IDs: UIACGF
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Intracranial Aneurysm
Keywords: cognitive function; quality of life; anxiety; depression; neurological function
MeSH Terms: conditions — Intracranial Aneurysm; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective single-center cohort study aims to identify the incidence of cognitive dysfunction after unruptured aneurysm operation and explore the influencing factors. The primary end point is the cognitive dysfunction at 6 months after operation.The features of cognitive function, mental status, neurological function recovery, and quality of life of patients with unruptured intracranial aneurysms at different time points would be analyzed.

DETAILED DESCRIPTION:
This main topics is to identify and screen the patients with unruptured aneurysm who likely to suffer from cognitive dysfunction. All examinations were administered by a trained neuropsychologist.The assessment of cognitive function and mental state would be performed before operation and 6 months after operation, with the use of Montreal Cognitive Assessment Scale (MoCA) for the cognitive function, the Hamilton Anxiety Scale (HAMA) and the Hamilton Depression Scale (HDMA) tests for the mental state. The Cognitive dysfunction at 6 months after operation would be the primary end point, and the underlying factors responsible for the declined cognitive function would be analyze. The assessment of neurological function and quality of life would be performed before operation,3 months after operation and 6 months after operation, with the use of the Modified Rankin Scale(mRS) and the Functional Activities Questionnaire(FAQ) for the neurological function, the Richards-Campbell Sleep Questionnaire(RCSQ) and the 36-item short from health survey(SF-36) tests for the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. At least one imaging (CTA / MRI / DSA) study to confirm unruptured intracranial aneurysms for the patients who would undergo surgical treatment for the first time.;
2. Patients who live independent with minimal care support, mRS score ≤3 points;
3. Age > 14 years old;
4. Han ethnicity, Right handed, can complete the test;
5. Patient or family agrees to sign informed consent.

Exclusion Criteria:

1. Other cerebrovascular diseases，such as ischemic stroke, arteriovenous malformation, etc;
2. With an unexplained subarachnoid hemorrhage;
3. History of Neurological disease surgery;
4. Previous psychiatric and dementia history that cannot communicate with other people;
5. Patients who refused to follow up.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the patients with unruptured intracranial aneurysms who treated in neurosurgery at Xuanwu Hospital
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
the Incidence of cognitive dysfunction at 6 months after operation | the 6th month after operation of the patient inclusion in the study
  The Montreal Cognitive Assessment Scale (MoCA) scale contains 8 cognitive domain,11 items and is suitable for assess cognitive function which including: Attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation.. 1 point for each correct answer. No points if they make any errors. The total score is 30 points. For those who have been educated for 12 years or less and the total score of MoCA is less than 30, one point is added to the total MoCA score. According to the results of MoCA assessment, Patients were divided into two groups: cognitive dysfunction group and cognitive function normal group. MoCA score ≥26 points suggested normal cognitive function (CN).

SECONDARY OUTCOMES:
the difference in the percentage of patients with HAMA score ≥14 before operation and 6 months after operation | before operation and the 6th month after operation of the patient inclusion in the study
  The Hamilton Anxiety Scale (HAMA) scale contains 14 items and is suitable for the adults with anxiety. Each item is divided into 5 grades evaluated using 0 to 4 scores. The total scores of HAMA scale can reflect patients' anxious condition to some extent. The total scores of less than 7 is regarded as no anxiety, 7 or more possible anxiety, 14 or more definite anxiety, 21 or more marked anxiety, 29 or more severe anxiety. In this study, Anxiety is defined as≥14 points.
the difference in the percentage of patients with HDMA score ≥14 before operation and 6 months after operation | before operation and the 6th month after operation of the patient inclusion in the study
  The Hamilton Depression Scale (HAMD) scale contains 24 items and is suitable for the adults with depression. Each item is divided into 5 grades evaluated using 0 to 4 scores. The total scores of the HAMD scale can reflect patients' depressive condition to some extent. The total scores of less than 8 is regarded as no depression, 8 to 16 mild depression, 17 to 24 moderate depression, and more than 24 severe depression. In this study, Depression is defined as≥14 points.
the tendency of mRS scores and the difference in the percentage of patients with mRS scores 0-3 and 4-6 points before operation, 3 months after operation, and 6 months after operation | before operation ,the 3th month and the 6th month after operation of the patient inclusion in the study
  The Modified Rankin Scale (mRS) is a valid and clinically relevant instrument that is used to assess recovery (death, disability, and dependence) after stroke and is a commonly used outcome measure in SAH studies. The mRS ranges from 0 (no symptoms) to 6 (death). Unfavourable outcome in survivors is defined as mRS 3-5.
the tendency of SF-36 scores before operation, 3 months after operation, and 6 months after operation | before operation ,the 3th month and the 6th month after operation of the patient inclusion in the study
  36-item short form health survey(SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Master, Study Chair — Xuanwu Hospital, Beijing